CLINICAL TRIAL: NCT02398019
Title: Clinical Trial to Evaluate Facticity and Security for the Use of an Increased Adsorption Capacity Membrane (oXiris®) During Cardiopulmonary Bypass Surgery
Brief Title: Clinical Trial to Evaluate the Use of an Adsorption Membrane (oXiris®) During Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Gambro Renal Products, Inc. (Industry)
Responsible Party: Principal Investigator, JOSE LUIS PEREZ FERNANDEZ, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIRAKI 01-2014
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Surgical Procedures; Cardiopulmonary Bypass
Keywords: CPB; oXiris®; SIRS; AKI; Cytokines; CSA-AKI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPB-OXIRIS® (Experimental): Non emergent cardiac surgery patients with CPB requirement.
  Interventions: Device: OXIRIS®
- CPB-Standard (No Intervention): Non emergent cardiac surgery patients with CPB requirement.

INTERVENTIONS:
Device: OXIRIS® — OXIRIS® membrane set is composed of a 1.5 m2 copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface and adhered heparin during set´s fabrication [OXIRIS® (Baxter Gambro)].
  PrismafleX eXeed™ II (Hospal) with OXIRIS® set will then be connected to CPB circuit. Blood flow between 150-200 ml/min will be derivatised from the CPB circuit into the PrismafleX eXeed™ so that it all flows through OXIRIS® membrane. Flow, pressure and alarms will be controlled by PrismafleX eXeed™ independently from CPB circuit.
  OXIRIS® membrane will be only employed for adsorption (neither convection nor diffusion will be performed) during all CPB time.
  Arms: CPB-OXIRIS®

SUMMARY:
Patients whom require cardiopulmonary bypass (CPB) during surgery present systemic inflammatory response syndrome (SIRS) due to blood cell activation and cytokine release to circulation. SIRS can lead to organ dysfunction due to hemodynamic compromise (vasodilatation plus leak syndrome) and/or cytokine mediated cell injury. Renal dysfunction is a major adverse complication after CPB surgery. Investigators hypothesize that the use of an increased adsorption membrane (OXIRIS®) during CPB is safe and presents low technical complexity. The safe use of OXIRIS® will reduce cytokine circulatory levels therefore decreasing SIRS and its systemic effects specially those concerning renal function. Therefore, patients receiving (OXIRIS®) could potentially present less cardiac surgery-associated acute kidney injury (CSA-AKI), and lower intensive care unit (ICU) and hospital length of stay.

DETAILED DESCRIPTION:
The oXiris® set connection to CPB

* The PrismafleX eXeed™ II (Baxter) system control unit will be used to deliver CRRT and thus connected to the CPB circuit through the oXiris® set lines.
* Priming. For oXiris® set priming use 2 L of normal saline according to the software instructions.
* Connection. Using a three-way stopcock, oXiris® set must be connected to the arterial line just after the oxygenator to derive blood into the oXiris® set and then returned into the venous reservoir through the return line. No additional vascular access will be required to deliver treatments.
* Modality. The Slow Continuous Ultrafiltration modality (SCUF modality) must be selected with no pre-set ultrafiltration rate (ultrafiltration rate: 0 ml/hr). A blood flow between 200-300 mL/min was set in the PrismafleX eXeed™ II (blood was derived through the arterial positive pressure line just after the oxygenator) to be delivered into the oXiris® set and then returned into the venous reservoir through the return line.
* All treatments should be delivered after reaching full-flow CPB.
* CRRT flow, pressure and alarms will be controlled in the PrismafleX eXeed™ II screen, independently from CPB circuit.
* If CPB is stopped for any reason, then PrismafleX eXeed™ II should be stopped temporarily to avoid alarm warning and/or any harm to the patient.
* No additional anticoagulation method will be needed besides the systemic anticoagulation required for the cardiopulmonary bypass pumping.
* The return line clamp (blue clamp) should be adjusted to reach a slight positive return pressure in order to avoid low-pressure alarm warning.

PrismafleX eXeed™ II weaning instructions. 5-10 min before the end of CPB, start the blood-return procedure into the venous reservoir of the CPB using 1 L of normal saline. Connect the solution into the three-way stopcock. Subsequently, set PrismafleX eXeed™ II flow in 80-100 ml/min. Select STOP in the PrismafleX eXeed™ II screen. Adjust the three-way stopcock to allow saline to flow into the oXiris® set arterial line an restart PrismafleX eXeed™ II to return blood into the venous reservoir.

• Register all manoeuvres, changes and adjustments in software settings and any technical problem during the procedure.

The oXiris® membrane will be only employed for adsorption (neither convection nor diffusion will be performed) during all CPB time. Using CPB flow, patient will not require venous catheter access neither changes in CPB normal settings.

The oXiris® membrane set is composed of a 1.5 m2 copolymer of acrylonitrile and sodium methylsulfonate (AN 69) with polyethylenimine treated surface and adhered heparin during set´s fabrication [oXiris® (Baxter Gambro)].

All blood samples collected during study will be obtained from CPB circuit or central venous catheters (standard cardiac surgery protocol).

During all CPB time besides the ordinary cardiac surgery assistance team, a supplementary CRRT expert team will be present in those patients randomized to CPB-oXiris®.

Blood samples and all variables will be equally collected and registered in the control group (CPB-Standard) with no modifications from CPB standard practice.

Adverse events will be reported (in less than 24 hours if severe) to the sponsor centre to be properly evaluated. If the severe adverse event (SAE) is finally evaluated by the study board as related to the intervention arm, urgent notification to health authorities must proceed and study should be interrupted until further decision.

Investigators will warrant a correct protocol application. Study data will be reviewed by an external monitoring committee from the clinical assay research central unit (UCICEC - IDIBELL). Monitors will contrast registered data from the collection data form (CDF) with data from patients' medical record. All patients' medical records will be indefinitely saved in electronic format to be reviewed if necessary.

Efficacy Assessments:

1. Registered variables and follow-up. Renal function related parameters Plasma creatinine and urine output will be registered at baseline, prior to CPB, at ICU admission, 6 hours ,12 hours, 24h postCBP and every 24h during the first week after cardiac surgery in order to evaluate CS-AKI based on KDIGO AKI criteria (KDIGO criteria Kidney inter., Suppl. 2012; 2: 1-138.) Renal function will be checked at hospital discharge.

   Hemolysis parameters Cell-free serum hemoglobin levels will be determined in plasma. These determinations will be measured at times T1 (at the end of CPB), and T3 (24 hours after ICU admission).

   Inflammatory response parameters Interleukin-1β (IL-1β), tumor necrosis factor alpha (TNF-α), monocyte chemotactic protein-1 (MCP-1), interleukin-4 (IL-4), interleukin-6 (IL-6), interleukin-8 (IL-8), interleukin-10 (IL-10), interleukin-18 (IL-18), complement 5a (C5a), high mobility binding protein 1 (HMBP-1), RANTES, GRO-alpha, leukocytes count, lactate, and D-dimer levels will be determined in plasma.These determinations will be measured baseline (0 hours), and at times T1 (at the end of CPB), T2 (ICU admission) and T3 (24 hours after ICU admission).

   Ordinary laboratory parameters Plasmatic urea, potassium, albumin, magnesium, phosphate, glucose, sodium, chloride, AST, ALT, blood cell count and coagulation times will be determined following the ordinary cardiac surgery protocol (every 8 hours during the first 24h).

   Clinical and respiratory parameters Hemodynamic and respiratory parameters will be registered every hour. Arterial and venous blood gases with arterial lactate will be determined every 8 hours during the first 24 hours. Temperature, heart rate, arterial blood pressure (systolic, diastolic, and mean), central venous pressure, vasopressor and/or inotrope dose will be registered during surgery and at ICU according to standard protocol.

   Demographic and clinical record data Age, gender, weight, height, relevant clinical records, previous or chronic medication, type of cardiac surgery, surgery times, time on CPB, surgical complications, blood transfusions during and after surgery, prognostic scores (SOFA, APACHE II and SAPS II), ICU stay, hospital stay. Clinical outcome (survival at discharge, 28 and 90 days) and renal outcome (renal function, and RRT requirements).
2. Techniques

   Cell-free serum hemoglobin analysis

   Cell-free serum hemoglobin concentration will be measured using the Cayman's Hemoglobin Colorimetric Assay Kit (Cayman Chemical, Ann Arbor, Michigan). Blood samples will be obtained at T1 and T3 into VACUETTE® Serum tubes (Greiner Bio One GmbH, Kremsmünster, Austria). After clotting at room temperature, serum will be separated by centrifugation at 2000 g for 15 minutes and stored at -80°C in 1 mL aliquots until use.

   Cell-free serum hemoglobin concentrations will be determined using manufacturer's protocols with provided calibration standards. All samples will be processed in duplicate. Changes in absorbance at 560 nm will be measured using a 96-well plate reader.

   Cytokines analysis

   IL-1, IL-6, IL-8, IL-10, IL-18, TNFα, MCP-1, HMBP-1, RANTES, GROα quantification will be performed with multiplex new technology. MILLIPLEX (Millipore) magnetic balls system will be used.
3. Study Limitations

   SIRS harmful effects which are initiated during CPB may persist after surgery and this is an important limitation as our study only evaluates the use of increased adsorption membranes during CPB. However, investigators hypothesize that the important effect on cytokine levels during CPB will be observed. Furthermore, patients requiring non emergent cardiac surgery represent a non absolutely homogeneous cohort and this could introduce potential bias in main and secondary objectives. To avoid this potential bias, temporary sequential randomization has been performed and advanced chronic renal failure patients have been excluded.
4. Statistical analysis

Missing data will try to be avoided by an exhaustive patient´s follow up by study investigators. Data registry has been created to include all variables with written individual data collection forms (DCF). Data will be bedside registered by the study members but final software database registration will be done by the statistics outside investigator who has no contact with patients situation. Cytokines levels will be introduced in DCF when measured.

Statistical analysis will be done by the statistics investigator who wont have any role in patient´s selection, randomization, or follow up. SPSS v. 20.0 for statistical analysis will be used. Variable distribution will be studied and logarithmic transformation will be used on those variables that don't present normal distribution, presumably cytokine levels. Univariate analysis comparing clinical, demographic, biochemical, metabolic, hemodynamic and respiratory baseline variables between both arms (CPB-OXIRIS® and CPB-Standard), will be done with two-tailed t test for continuous variables and chi-square test for categorical variables. Variables determined several times (T0, T1, T2, T3) will be analysed using a one-way repeated measures ANOVA test in order to demonstrate differences between both arms. Multivariate analysis will be completed to control those clinically relevant confounding variables as well as to discover baseline differences. Arm intervention (CPB-OXIRIS®, CPB-Standard) will be considered as the main independent variable adding other control independent variables. Intervention safety will be measured by the presence of any adverse effects not related to the standard technique. This effects will be recorded during CPB, after CPB, and during the first 24 hours postsurgery.

As the study is measuring cytokine levels in four different moments (T0, T1, T2, T3), in order to maximize statistical power and reduce control variables number, the area under the curve (AUC) we´ll be determined for every cytokine during the first 24 hours. Due to this statistical maneuver investigators will obtain a continuous variable that represents each cytokine level during the biochemical study period (24 hours). To evaluate if the arm intervention improvement in terms of efficacy and safety could be related to cytokine levels during the first 24 hours, a mediation complementary analysis will be done considering cytokine (represented by AUC) as a mediator between the independent variable (intervention arm) and the effect we study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 18 years old.
* Non emergent cardiac surgery requiring CPB.
* Written informed consent from patient or legal surrogates

Exclusion Criteria:

* Missing informed consent.
* Planned CPB hypothermia <32ºC or cardiac arrest.
* Emergency surgery.
* Acute infective endocarditis.
* Immunosuppressive treatment or steroids (prednisone > 0.5 mg/kg/day or equivalent).
* Autoimmune disorder.
* Transplant receptor.
* Advanced Chronic Kidney Disease (CKD 4 or 5).
* Renal replacement therapy (RRT) in the last 90 days.
* Documented intolerance to study device.
* Inclusion in other ongoing study within the last 30 days.
* Pregnancy.
* Coexisting illness with a high probability of death (inferior to 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety with the use of CPB. Number of complications reported. | 24 hours
  Patients who underwent cardiac surgery with no related complications due to CPB (0 complications). Complications will be defined as those adverse effects related to technique that need an extra attention out of standard proceedings.
Cell-free serum hemoglobin | 24 hours
  Cell-free serum hemoglobin concentration will be measured in order to evaluate intravascular hemolysis.
  Determinations will be measured at T1 (CPB end), and T3 (24hours).

SECONDARY OUTCOMES:
Cytokine circulatory levels during CPB and up to 24 hours after surgery. | 24 hours
  Cytokine circulatory levels during CPB and up to 24 hours after surgery. Cytokine removal: interleukin-1β (IL-1β), tumor necrosis factor α (TNF-α), interleukin-4 (IL-4), interleukin-6 (IL-6), and interleukin-10 (IL-10) levels will be determined in plasma.
  Determinations will be measured baseline (0hours), and at T1 (CPB end), T2 (ICU admission), and T3 (24hours).
Creatinine and Urine output after cardiac surgery. | 7 days
  Renal function in terms of creatinine and urine output will be registered every 24h after cardiac surgery up to the first week.

CONTACTS AND LOCATIONS:
Overall Officials: Xose Luis Perez Fernandez, MD, Principal Investigator — Hospital Universitari de Bellvitge; Joan Sabater Riera, MD Ph.D, Study Director — Hospital Universitari de Bellvitge; Paola Cárdenas, MD, Study Chair — Hospital Universitari de Bellvitge; Enric Boza, MD, Principal Investigator — Hospital Universitari de Bellvitge; Erika Plata-Menchaca, MD, Principal Investigator — Institut d'Investigació Biomèdica de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain